CLINICAL TRIAL: NCT05428709
Title: Women In Steady Exercise Research - Window of Opportunity for Exercise and Tumor Biology
Acronym: WISER-WIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving academia
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen Sturgeon, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00019979
Record Dates: First submitted 2022-04-22; First posted 2022-06-23 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: acute exercise; ctDNA; exerkines; tumor perfusion; oxygen saturation
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute exercise (Experimental): Participants will be asked to walk or jog on a treadmill for a maximal exercise test.
  Interventions: Behavioral: Acute Exercise

INTERVENTIONS:
Behavioral: Acute Exercise — Participants will be asked to walk or jog on a treadmill for a maximal exercise test.

SUMMARY:
The primary aim is to examine changes in tumor perfusion, oxygen saturation, and tumor physiology before and following acute physical activity in breast cancer patients.

The secondary aim is to examine changes in circulating tumor DNA (ctDNA) levels before and following acute physical activity in breast cancer patients.

The tertiary aim is to explore changes in circulating exerkines (cytokines and growth factors altered by exercise) before and following acute physical activity in breast cancer patients.

DETAILED DESCRIPTION:
The proposed study seeks to leverage acute exercise physiology as a tool to better understand multiple clinical and mechanistic issues in exercise oncology. An acute exercise bout causes functional changes such as increases in heart rate and stroke volume leading to increased cardiac output and increased systemic blood flow. These systemic effects also increase tumor blood flow (perfusion). Additionally, an increase in mean arterial pressure increases oxygen diffusion distance within the tumor. Further, acute exercise mobilizes NK cells, cytokine signaling, and a myriad of other molecular and cellular transducers of exercise. Our study of acute exercise physiology in breast cancer patients will address several significant knowledge gaps both clinically and mechanistically.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer patients
* Breast tumor is more than 2 cm (T2)
* With or without lymph node involvement (N0-3)
* With or without metastases (M0-M1)
* No initiation of neoadjuvant treatment
* Pre-surgical breast resection

Exclusion Criteria:

* Current use of anticoagulants, including Vitamin K antagonists (e.g. Warfarin), Direct Oral Anticoagulants (DOACs) (e.g. Pradaxa, Eliquis, Xarelto, Bevyxxa, Savaysa), low molecular weight heparins (LMWH), Fragmin, Lovenox, heparin.
* Body weight <100 lbs
* Tis, T0, T1
* Started neoadjuvant therapy
* Absolute contraindications for exercise stress testing by self-report:

  * acute myocardial infarction (3-5 days)
  * unstable angina
  * uncontrolled arrhythmias causing symptoms or hemodynamic compromise
  * syncope
  * acute endocarditis
  * acute myocarditis or pericarditis
  * uncontrolled heart failure
  * acute pulmonary embolus or pulmonary infarction
  * thrombosis of lower extremities
  * suspected dissecting aneurysm
  * uncontrolled asthma
  * pulmonary edema
  * room air desaturation at rest ≤85%
  * respiratory failure
  * acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
  * mental impairment leading to inability to cooperate
  * decisional impairment
* Non-English speaking
* Pregnant women
* Children

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Changes in total hemoglobin | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  Total hemoglobin will be quantified using photoacoustic imaging and the % difference will be determined 1) before cardiopulmonary exercise (CPET) (Time 0), 2) immediately after CPET (Time 1), 3) 30 min after CPET (Time 2) , and 4) 2 hours after CPET (Time 3).
Changes in oxy-hemoglobin | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  Oxy-hemoglobin will be quantified using photoacoustic imaging and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.
Changes in deoxy-hemoglobin | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  Deoxy-hemoglobin will be quantified using photoacoustic imaging and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.
Changes in oxygen saturation | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  Oxygen saturation will be quantified using photoacoustic imaging and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.

SECONDARY OUTCOMES:
Changes in ctDNA level | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  ctDNA level will be measured in blood and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.
Exerkine: TGF-β | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  TGF-β will be measured in blood and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.
Exerkine: VEGF-A | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  VEGF-A will be measured in blood and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.
Exerkine: S1P | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  S1P will be measured in blood and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.
Exerkine: TSP-1 | baseline or before cardiopulmonary exercise (CPET), immediately after CPET (an average of 12 min following baseline), 30 min following CPET, and 2 hours following CPET
  TSP-1 will be measured in blood and the % difference will be determined at Time 0, Time 1, Time 2, and Time 3.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Sturgeon, PhD, MEd, MS, Principal Investigator — Penn state University College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States